CLINICAL TRIAL: NCT04141293
Title: Hemodynamic Effects of Changes in Transpulmonary Pressure During Recruitment Maneuver in Patients Under Pressure Support Mechanical Ventilation
Brief Title: Hemodynamic Effects of Changes in Transpulmonary Pressure During Recruitment Maneuver in Patients Under Pressure Supported Mechanical Ventilation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical problems and employee shortage
Sponsor: Kiskunhalas Semmelweis Hospital the Teaching Hospital of the University of Szeged (Other Government)
Responsible Party: Principal Investigator, András Lovas, Head of Department, Kiskunhalas Semmelweis Hospital the Teaching Hospital of the University of Szeged
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 101/2017-SZTE
Record Dates: First submitted 2017-08-30; First posted 2019-10-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible patients (Experimental)
  Interventions: Procedure: alveolar recruitment

INTERVENTIONS:
Procedure: alveolar recruitment — Alveolar recruitment is a procedure to re-expand collapsed lung regions with the transient increment in transpulmonary pressure.

SUMMARY:
According to the anatomical proximity of the heart temporarily elevated intrathoracic pressures may have direct and indirect effects on the cardiovascular system. Undesirable hemodynamic effects of a recruitment maneuver primarily arise from the transiently increased airway pressure, manifesting in decreased right heart filling, increased pulmonary vascular resistance, a drop in left ventricular systolic transmural pressure, right and left heart ventricular interactions and subsequent changes in cardiac index. These effects can be more pronounced in patients suffering from ARDS, a condition commonly accompanied by hemodynamic instability. The complex pathophysiological changes account for why routine intensive care monitoring, such as invasive arterial blood pressure or central venous pressure monitoring is insufficient to follow hemodynamic changes under recruitment maneuver.

Previous studies by the same research team confirmed that the alveolar recruitment maneuver improves oxygenation in patients with moderate-to-severe hypoxemic respiratory failure under pressure supported ventilation. Following recruitment maneuver, arterial oxygenation increased in 74 % of all patients. However, there is lack of information regarding the actual degree of changes in transpulmonary pressure and the consequent hemodynamic alterations.

The primary aim of the study is to evaluate precisely the transpulmonary pressure changes during recruitment in patients with severe hypoxemic respiratory failure ventilated in pressure support mode following insertion of a balloon-catheter into the esophagus. In the meantime, hemodynamic changes are monitored by PiCCO and transthoracic echocardiography, and lung field aeration by electric impedance tomography.

ELIGIBILITY:
Inclusion Criteria:

* orotracheal intubation
* pressure supported ventilation
* moderate-to-severe hypoxemic respiratory failure according to ARDS Berlin Criteria Moderate: 100 Hgmm ≤ PaO2/FiO2 ≤ 200 Hgmm, PEEP ≥ 5 cmH2O Severe: PaO2/FiO2 ≤ 100 Hgmm, PEEP ≥ 5 cmH2O

Exclusion Criteria:

* age < 18 years
* pregnancy
* previous pulmonary resection, pulmonectomy
* clinically verified, end-stage COPD
* severe hemodynamic instability (i.e. refractory shock to vasopressors)
* severe emphysema and/or spontaneous pneumothorax in past medical history
* contraindications of a balloon-catheter (e.g. esophageal abscess, esophageal perforation, esophageal diverticulosis, esophagus tumor, esophagus varix, recent esophagus or gastric surgery, severe coagulopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of transpulmonary pressure and hemodynamic changes during alveolar recruitment | Approximately 35 minutes
  Changes in transpulmonary pressure during alveolar recruitment will be compared to the subsequent hemodynamic alterations

SECONDARY OUTCOMES:
Changes in left and right ventricular volume (systolic ventricular interdependence) | Approximately 3 minutes
  Left ventricular end-systolic eccentricity index will be assessed by transthoracal echocardiogarphy and will be compared with transpulmonary pressure alterations.
Changes in pulmonary air content | Approximately 30 miniutes
  Changes in pulmonary atelectasis will be assessed by electrical impedance tomography (EIT) - mean impedance variation in % and will be compared with arterial oxygen content.
Changes in arterial oxygen content | Approximately 5 minutes
  Pre- and post-recruitment arterial oxygenation (PaO2 mmHg) will be measured by blood gas machine and will be compared to EIT measurements.
Changes in hemodynamic parameters (SV) | 35 minutes
  Changes in stroke volume (ml)
Changes in hemodynamic parameters (MAP) | 35 minutes
  Changes in mean arterial pressure (mmHg)
Changes in hemodynamic parameters (HR) | 35 minutes
  Changes in heart rate (1/min)
Changes in hemodynamic parameters (CI) | 35 minutes
  Changes in cardiac index (l/min/2m)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Department of Anesthesiology and Intensive Therapy, Szeged, Csongrád megye, Hungary

REFERENCES:
- [Background] Lovas A, Szakmany T. Haemodynamic Effects of Lung Recruitment Manoeuvres. Biomed Res Int. 2015;2015:478970. doi: 10.1155/2015/478970. Epub 2015 Nov 22. PMID 26682219
- [Background] Lovas A, Nemeth MF, Trasy D, Molnar Z. Lung recruitment can improve oxygenation in patients ventilated in continuous positive airway pressure/pressure support mode. Front Med (Lausanne). 2015 Apr 21;2:25. doi: 10.3389/fmed.2015.00025. eCollection 2015. PMID 25954744
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2014 Mar 6;370(10):980. doi: 10.1056/NEJMc1400293. No abstract available. PMID 24597883
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452